CLINICAL TRIAL: NCT00776958
Title: Multi - Center Database/Registry of Subjects at High Risk for Ovarian or Breast Cancer - A Lynne Cohen Consortium Project
Brief Title: Lynne Cohen Consortium Project: Multi-Center Database/Registry
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Lynne Cohen Foundation for Ovarian Cancer Research (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0067
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Ovarian Cancer; Breast Cancer
Keywords: A Lynne Cohen Consortium Project; Multi-Center Database Registry; High Risk; Cancer; Breast; BRCA1 or BRCA2 gene; Ovary; Questionnaire
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Neoplasms; Fanconi Anemia, Complementation Group D1 | interventions — Surveys and Questionnaires; Demography; Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ovarian or Breast Cancer Study Registry
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Information Collection for Entry into Multicenter Registry: Survey 5-10 minutes. Participation lasts as long as patient agrees to continue having study information collected
  Other Names: Survey; Demographics; Data Collection

SUMMARY:
Goals of this registry:

1.1 To collect and store very limited demographic information (age, birthdate, race and ethnicity), limited cancer risk and breast and ovarian disease history, as well as limited family history of breast and ovarian cancer on patients who are at risk of breast or ovarian cancer or who have had a diagnosis of either cancer,

1.2 To make available summary information (in an anonymous form) regarding the subjects in this registry to Consortium members, and other investigators, who can use these data to plan research projects and evaluate the feasibility of such projects,

1.3 To make available summary information (number of new patients seen in the clinic, number of mutations, number of preventive surgeries, average age of patients seen) to the Lynne Cohen Foundation for Ovarian Cancer Research, in order to document the numbers of subjects who utilize their supported clinics.

DETAILED DESCRIPTION:
Information Collection for Entry into Multicenter Registry:

If you agree to take part in this study, a study staff member will collect the following information by asking you at a clinic visit and checking your medical records. The following information will be entered in the registry:

your demographic information (your sex, year of birth, and race/ethnicity) whether any member of your family has a history of ovarian and/or breast cancer whether any member of your family has any known genetic markers that may mean a higher risk of developing a cancer a brief summary of your history of breast and/or ovarian disease and whether you have any known genetic markers that may mean a higher risk of developing breast and/or ovarian cancer a brief summary of the results of the clinic visit on the day you agreed to take part in this study (Day 1)

Follow-Up Information Collection:

Each time you visit the M. D. Anderson high-risk clinic (either the high-risk breast cancer clinic or the high-risk ovarian cancer clinic), the study staff will check your medical records and enter in the registry any updates to your cancer risk information. You will also be asked if any family members have been diagnosed with ovarian and/or breast cancer, and this will be entered in the registry.

If you miss any of your planned clinic visits, the study staff may contact you by phone to collect this information, contact you by mail to send you a questionnaire with this information, and/or reschedule your appointment. If you receive a questionnaire by mail, you will fill it out and mail it back to the research staff in the stamped, self-addressed envelope that will be provided to you. It should take about 5-10 minutes to complete.

Study Data:

The study staff plans to keep all personal identifying information (such as your name) strictly confidential. Your data will be handwritten on paper forms that will be stored in a locked file cabinet. The study staff will enter your data into the multicenter database (registry) with your participant identification (ID) number but not your name or other identifying information. The registry is password-protected. Only designated members of the study staff will have access to the participant ID numbers and be able to link the data to you. This is to allow medical information related to your data to be updated as needed. The linking information will be saved securely (on a password-protected computer) in the research office.

The multicenter registry is called the Lynne Cohen registry. It is maintained at the University of Southern California Norris Comprehensive Cancer Center.

Use of Registry for Planning Future Research:

Lynne Cohen clinics make up the multicenter group of clinics that are involved in this study. If a researcher at any Lynne Cohen clinic is planning to perform a research study involving ovarian or breast cancer causes or prevention, he or she can contact the Lynne Cohen Foundation. A staff member at the Lynne Cohen Foundation will check to see how many patients are included in the registry. This will help the researcher find out how many people the researcher may be able to ask to join his or her study. That number of people will also help the researcher decide if the planned study is feasible. The number of patients in the registry is the only information that will be shared with these researchers.

Length of Study Participation:

Your participation in this study will last for as long as you agree to keep having this study information collected.

When your participation in this study ends, the M. D. Anderson study staff will delete or destroy any personal identifying information and contact information collected. The rest of the study data will continue being stored in the registry.

This is an investigational study.

Up to 1000 patients will be enrolled in this multicenter study. Up to 200 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Women who are 18 or older and meet one or more of the following criteria.
2. Personal history of breast and/or ovarian cancer.
3. Family history of breast and/or ovarian cancer (one or more relatives).
4. Carrier of a mutation in the BRCA1 or BRCA 2 gene, or the presence of one of these mutations in a family member.

Exclusion Criteria:

1) None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women seen at a member clinic of the Lynne Cohen Consortium having, or at high risk of either ovarian or breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2008-07; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Collection of Demographic and Cancer Risk Information on Women Who Are at High Risk for Ovarian or Breast Cancer | 9 Years

SECONDARY OUTCOMES:
Establish Repository of Minimal Basic Data (Multicenter Registry) | 9 Years

CONTACTS AND LOCATIONS:
Overall Officials: Karen H. Lu, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (4):
- United States (4):
  - University of Alabama, Birmingham/Department of OB/GYN, Birmingham, Alabama
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - NYU Cancer Institute, New York, New York
  - UT MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org